CLINICAL TRIAL: NCT03785938
Title: Mucositis and Infection Reduction With Liquid Probiotics in Children With Cancer: a Randomised-controlled Feasibility Study
Brief Title: Mucositis and Infection Reduction With Liquid Probiotics in Children With Cancer
Acronym: MaCROS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Hadeel Hassan, Clinical Research Fellow, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: IRAS PROJECT ID: 246313
Record Dates: First submitted 2018-12-05; First posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Pediatric Cancer
Keywords: pediatric; cancer; malignant haematology; transplant; probiotics; mucositis; infection; supportive care
MeSH Terms: conditions — Neoplasms; Mucositis; Infections | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Double blinded randomised-controlled feasibility study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The liquid probiotic/placebo will be blinded by the pharmacy team and LTHT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Participants will start the course of liquid probiotic on the first day of their course of chemotherapy. This can be taken orally, or using an nasogastric or gastrostomy tube and will continue this for 14 days. Doses will be adjusted according to the age of the participant as follows:
  1-4 years:20ml once a day 4-11 years: 0.5ml/kg once a day 12-18 years: 1ml/kg once a day
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Participants will start the course placebo on the first day of their course of chemotherapy. This can be taken orally or using an nasogastric or gastrostomy tube and will continue this for 14 days. Doses will be adjusted according to the age of the participant as follows:
  1-4 years:20ml once a day 4-11 years: 0.5ml/kg once a day 12-18 years: 1ml/kg once a day
  Placebo will be delivered in similar, packaging, appearance and taste.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Liquid probiotic supplied by the company Symprove
  Other Names: Symprove liquid probiotic
  Arms: Probiotic
Other: Placebo — Placebo made of maltdextrin. Will be similar in taste and consistency
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the feasibility of an randomised-controlled trial to investigate the efficacy of liquid probiotics to prevent or reduce mucositis and infection in children diagnosed with cancer who are undergoing treatment with regimes likely to cause mucositis.

DETAILED DESCRIPTION:
TRIAL DESIGN

This will be a single-centre double-blind randomised-controlled feasibility study.

TRIAL SETTING

This study will take place at Leeds Teaching Hospital Trust (LTHT), Leeds UK. Participants will be approached whilst admitted as inpatients (typically the paediatric haematology oncology wards) and during outpatient clinics.

METHOD

Allocation sequence from a randomisation schedule will be generated A screening or trial ID number will be assigned to each participant.

The allocation sequence will be concealed from health care professionals, participants and families. Only the pharmacy team involved in randomisation, allocation will not be blinded to allocation sequence and generation.

Following identification, confirmation of eligibility, consent and allocation of trial ID of the participant, a prescription will be produced and the probiotic or placebo will be allocated accordingly.

Appearance of the intervention and placebo will be similar in appearance, smell and taste. The placebo will include maltdextrin (a polysaccharide). Both the probiotic and placebo will be produced by the company Symprove.

Participants will start the course of probiotic or placebo on the first day of their course of chemotherapy orally, or using an nasogastric or gastrostomy tube and will continue this for 14 days. Doses will be adjusted according to the age of the participant as follows:

1-4 years:20ml once a day 4-11 years: 0.5ml/kg once a day 12-18 years: 1ml/kg once a day Placebo will be delivered in similar, packaging, appearance and taste.

Participants or their parents will be asked to fill in a diary (paper or electronic using a web-app) daily for 21 days in total. The diary will include questions to assess nausea, vomiting, diarrhoea, pain and oral mucositis. An example of the patient diaries offered is supplied. Either the participant or parent will fill in the diary on a daily basis for a minimum of 21 days.

The web-app is an electronic version of the paper diary. Participants will to chose their preferred method. Participants will be given the URL which they can download onto their phone as a web-app. Data provided by participants in the web-app will only be identified by their unique identification number and information will be transferred to an excel spread sheet.

Clinical records including electronic and written records will be reviewed to investigate any febrile episodes and infections for incidence and duration of fever/infection and duration of hospital stay until afebrile for 48 hrs. Any data collected from clinical records will be stored on an excel web sheet which will be kept on an NHS computer. Data on the excel spreadsheet will be identified using their unique identification number. Data will be collected and analysed on an NHS computer. The person collecting the data (the principal investigator) is also a member of the health care team and has access to clinical records as part of routine care.

Participants will be invited to participate in an optional interview exploring their experiences in taking part in the study. This will take up to 45 minutes and can be done over the phone or in person whilst in the hospital. The interviews will be recorded using an encrypted digital audio recorder.

Participants who chose to decline will also be invited to a short optional interview exploring why they chose to decline. This will approximately be a 10 minute discussion which will take place when the participant/their parent disclose they have decided to decline and will only take place if both the participant/parent and interviewer (the chief investigator) is present in the hospital.

ELIGIBILITY:
Inclusion Criteria:

Patients between the ages of 1 and 18 treated on paediatric cancer protocols receiving chemotherapy on regimens likely to cause mucositis.

Exclusion Criteria:

Patients who have already started the course of chemotherapy. Patients receiving radiotherapy or surgery alone. Patients diagnosed with an immunodeficiency (excluding IgA). Patients who have previously taken probiotics within the month prior to commencing the course of chemotherapy.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-20 (Estimated); Primary Completion 2019-07-20 (Estimated); Study Completion 2019-08-20 (Estimated)

PRIMARY OUTCOMES:
Recruitment | 6 months
  Proportion of eligible participants successfully recruited to the MaCROS study
Recruitment | 6 months
  Proportion and number of eligible participants successfully recruited to the MaCROS study
Compliance of taking the probiotic/placebo | 6 months
  Proportion of participants who are able to complete the 14 day course
Compliance of filling in the paper/web-app diary | 6 months
  Proportion of participants who are able to fill in and return the diary for 21 days
Cost-benefit evaluation of the study | 6 months
  Cost-benefit analysis of undertaking the study

SECONDARY OUTCOMES:
Incidence of mucositis in both groups | 6 months
  Proportion of participants who develop mucositis in both groups.
Comparison of mucositis in both groups | 6 months
  Mean difference of mucositis (if possible) between both groups
Proportion of participants who develop fever | 6
  Proportion of participants who develop fever Mean difference of fever (if possible) between both groups
Evaluate responsible guardian/participants experience of the MaCROS study | 6 months
  This optional part of the study will be done by undertaking recorded telephone or face to face interview

CONTACTS AND LOCATIONS:
Overall Officials: Hadeel Hassan, MBCHB MSc, Principal Investigator — University of Leeds

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hassan H, Kinsey S, Phillips B. Mucositis reduction with probiotics in children with cancer: a randomised-controlled feasibility study. Arch Dis Child. 2022 Mar;107(3):259-264. doi: 10.1136/archdischild-2020-319968. Epub 2021 Jun 30. PMID 34193407